CLINICAL TRIAL: NCT06875063
Title: The Safety, Tolerability, Efficacy, and Pharmacokinetic Characteristics of GB5005 Chimeric Antigen Receptor T-cell Injection in Treating Patients With CD19-positive Relapsed/Refractory B-cell Non-Hodgkin Lymphoma (B-NHL).
Brief Title: GB5005 CART-cell Injection in the Treatment of Patients With CD19-positive RR B-NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-17
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Non-hodgkin Lymphoma,B Cell; Relapsed Non-Hodgkin Lymphoma; Refractory Lymphoma; Chimeric Antigen Receptor T-cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose group (Experimental): GB5005 chimeric antigen receptor T-cell injection（1 × 10 ^ 6 cells/kg）
  Interventions: Drug: GB5005 CART
- Median dose group (Experimental): GB5005 chimeric antigen receptor T-cell injection（2 × 10 ^ 6 cells/kg）
  Interventions: Drug: GB5005 CART
- Medium to high dose group (Experimental): GB5005 chimeric antigen receptor T-cell injection（3 × 10 ^ 6 cells/kg）
  Interventions: Drug: GB5005 CART
- High dose group (Experimental): GB5005 chimeric antigen receptor T-cell injection（5 × 10 ^ 6 cells/kg）
  Interventions: Drug: GB5005 CART

INTERVENTIONS:
Drug: GB5005 CART — Included patients will receive GB5005 chimeric antigen receptor T-cell injection: A sterile syringe will be used to draw the assigned dose volume (calculated based on the patient's weight and converted to volume). The cells will be slowly infused intravenously at a rate of about 10 mL/min.
  Other Names: GB5005 chimeric antigen receptor T-cell injection

SUMMARY:
To evaluate the safety and tolerability of GB5005 in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma (B-NHL).

DETAILED DESCRIPTION:
Primary objectives: To evaluate the safety and tolerability of GB5005 in patients with CD19-positive relapsed/refractory B-cell non-Hodgkin lymphoma (B-NHL).

Secondary objectives: To assess the preliminary efficacy of GB5005 in patients with CD19-positive B-NHL; To describe the pharmacokinetic profile of GB5005 and observe its proliferation and persistence in the body; To explore the correlation between the pharmacokinetic characteristics of GB5005 and cytokine release syndrome (CRS) as well as neurological events.

ELIGIBILITY:
Inclusion Criteria:

1. The candidate is able to communicate effectively with researchers and sign informed consent forms in writing;
2. Age greater than or equal to 18 years old and less than or equal to 70 years old, regardless of gender; Sign informed consent form;
3. Non Hodgkin lymphoma confirmed by cytology and genetics;
4. Positive expression of CD19 in tumor cells confirmed by flow cytometry or pathological histology;
5. When screening, it meets the definition of recurrence or refractory: having received at least second-line or above systemic anti-tumor therapy (including autologous hematopoietic stem cell transplantation) containing rituximab (or other CD20 targeted drugs) and anthracycline drugs in the past, and disease progression (PD) or recurrence after the last treatment; Or recurrent patients who do not fully meet the above conditions but refuse chemotherapy and strongly demand CAR-T treatment;
6. There is no obvious evidence of central nervous system lymphoma on brain MRI;
7. Blood routine: Neutrophils ≥ 1.0 × 10 ^ 9/L; Hemoglobin ≥ 70 g/L; Platelets ≥ 50 × 10 ^ 9/L;
8. Coagulation function: fibrinogen ≥ 1.0 g/L; Activated partial thromboplastin time (APTT) ≤ ULN+10 s, prothrombin time (PT) ≤ ULN+3 s;
9. Liver and kidney function indicators: total bilirubin ≤ 1.5 times the upper limit of normal range (excluding Gilbert syndrome or hemolysis), ALT and AST ≤ 3.0 times the upper limit of normal range (ULN), serum creatinine ≤ 2.0 times the upper limit of normal range. If the above abnormalities are considered to be caused by tumor infiltration, they can be excluded;
10. Assessment of left ventricular ejection fraction (LVEF) ≥ 45% using echocardiography (ECHO) or radionuclide active vascular scanning (MUGA). (After corrective treatment and meeting the criteria, it can be included in the group);
11. Pulmonary function: Dyspnea ≤ CTCAE level 1 and SaO2 ≥ 92% in indoor air environment; 12. The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) in the United States ranges from 0 to 2 points;
12. Expected survival is greater than 6 months; 14. The subjects have sufficient levels of functional organs during screening;
13. Female participants of childbearing age must undergo a serum pregnancy test during screening and before receiving pre-treatment chemotherapy, and the result must be negative. They are willing to use highly effective and reliable methods of contraception within one year after using the study treatment;
14. Male participants who engage in active sexual activity with women with reproductive potential must be willing to use highly effective and reliable methods of contraception within one year after using the study treatment. Moreover, all males are strictly prohibited from donating sperm within one year after receiving research treatment infusion during the study period.

Exclusion Criteria:

1. Patients with a history of allergies to serum albumin and DMSO in the past;
2. Active hepatitis B virus (HBV) (HBV-DNA positive), hepatitis C virus antibody (HCV) (HCV-RNA positive), or human immunodeficiency virus (HIV) infection;
3. Within the past 2 years, terminal organ damage caused by autoimmune diseases such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, or the need for systemic use of immunosuppressive or other systemic disease control drugs;
4. History of unstable angina, myocardial infarction, coronary angioplasty, or significant heart disease within one year of enrollment;
5. Primary central nervous system tumors or hematological tumors with central nervous system metastases;
6. Uncontrolled mental illness;
7. Merge other life-threatening severe organ failure;
8. Participated in other clinical studies within 4 weeks;
9. Received live vaccination within 4 weeks of enrollment;
10. Using prohibited drugs: a. Hormones: Corticosteroids (defined as>20mg/day prednisone or equivalent) used at therapeutic doses within 7 days prior to leukocyte collection. But the use of physiological substitutes, local and inhaled steroids is allowed. b. Chemotherapy: rescue chemotherapy, including tyrosine kinase inhibitors (TKIs), received within 1 week before leukocyte collection. c. Donor lymphocyte infusion (DLI) received within 4 weeks before leukocyte collection. d. graft-versus-host disease (GvHD) treatment: systemic anti GVHD treatment received within 3 months before GB5005 cell infusion. e. Alenumab used within 6 months before leukocyte collection, or chlorofarabin or cladribin used within 3 months. f. Checkpoint inhibitors or stimulants used before enrollment (excluding those with more than 3 biological half lives);
11. Patients with known history of lung injury or hemorrhagic cystitis associated with cyclophosphamide treatment;
12. Women who are already pregnant, preparing for pregnancy during the trial period, or breastfeeding;

13：As per the investigator's judgment, the subject is unlikely to complete all required visits or procedures stipulated in the protocol (including the follow-up period) or has insufficient compliance with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) | Up to 3 months
  Complete remission rate was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Recurrence free survival time (RFS) | Up to 24 months
  Recurrence free survival time was defined as the time from the date of treatment initiation to the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first.
  PFS was defined as the time from the date of treatment initiation to the date of first documentation of definitive disease recurrence or date of death from any cause, whichever occurs first.
  PFS was defined as the time from the date of treatment initiation to the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first.
Overall survival（OS） | Up to 24 months
  Overall survival will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No